CLINICAL TRIAL: NCT04791176
Title: Phase II Study of Concurrent Lenvatinib and Intensity-modulated Radiotherapy (IMRT) for Advanced Hepatocellular Carcinoma
Brief Title: Phase II Study of Concurrent Lenvatinib and Radiotherapy for Advanced HCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, BO CHEN, Associate Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2508
Record Dates: First submitted 2021-03-06; First posted 2021-03-10 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma; Radiotherapy; Lenvatinib
Keywords: hepatocellular carcinoma; intensity-modulated radiotherapy; portal vein thrombosis; lymph node metastasis; Lenvatinib
MeSH Terms: conditions — Carcinoma, Hepatocellular; Lymphatic Metastasis | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lenvatinib and IMRT (Experimental): Concurrent Lenvatinib and IMRT, followed Lenvatinib maintenance for advanced hepatocellular carcinoma with portal vein or hepatic vein tumor thrombosis or lymph node involved
  Interventions: Radiation: concurrent lenvatinib and Radiotherapy, followed lenvatinib maintenance

INTERVENTIONS:
Radiation: concurrent lenvatinib and Radiotherapy, followed lenvatinib maintenance — Radiotherapy with IMRT or VMAT with 40-60Gy/20-30f; Concurrent Lenvatinib 12mg/day (for patients≥60 kg) or 8 mg/day (for patients<60kg ) qd po. (Note: Levatinib can be given to patients in four weeks before Radiotherapy is applied, so that it can control disease during waiting for Radiotherapy). Maintenance Lenvatinib 12mg/day (for patients≥60 kg) or 8 mg/day (for patients<60kg ) qd po until disease progress or unacceptable adverse events; six months is recommended but not mandatory.

SUMMARY:
This is a single-arm, open-label study performed at our hospital, patients with progression hepatocellular carcinoma (HCC) met inclusion criteria will be enrolled. Patients received oral lenvatinib 12mg/day (for patients≥60 kg) or 8 mg/day (for patients<60kg ) before local radiotherapy 4 weeks, large lesions were treated with IMRT for 40-60gy / 20-30f. Combined therapy will be taken until unacceptable treatment-related toxicities occurred or disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Patients had an HCC diagnosis confirmed either histologically or clinically according to the Chinese Society of Clinical Oncology guidelines for primary liver cancer 2019 version；
2. Aged ≥18 years and <80 years；
3. ECOG 0-1;
4. Live-GTV volume > 700ml;
5. BCLC stage C, HCC with portal vein or hepatic vein tumor thrombosis or lymph node involved (LN involved can be included one treatment planning);
6. Estimated life expectancy should be more than 3 months;
7. Patients with lung and / or bone metastases can be enrolled if those metastases couldn't effect the patients' life and quality of life within 3 months;
8. Child-Pugh Score A5,A6,B7;
9. Liver function: ALT is less than 1.5 times of the upper limit of normal; ALT is less than 0.5 times of the upper limit of normal, AST can be less than 6 times of the upper limit of normal, excluding the elevation of AST caused by heart infarction; ALT is 0.5 to 1.5 times of the upper limit of normal, AST is less than 1.5 times of the upper limit of normal;
10. ECG examination showed no obvious abnormality, no obvious cardiac dysfunction;
11. Renal function: CRE and BUN were within 1.5 times of the upper limit of normal value;
12. Blood routine: HB ≥ 80g / L, ANC ≥ 1.0 × 109 / L, PLT ≥ 40 × 109 / L;
13. Coagulation function: no bleeding tendency;
14. Informed and voluntarily participated in the study and signed informed consent.

Exclusion Criteria:

1. Currently in the process of other clinical trials within recently four weeks;
2. Previous abdominal radiotherapy and liver transplantation;
3. Patients with severe chronic diseases of heart, kidney, liver and other important organs;
4. Pregnant or lactating women;
5. Suspected or indeed drug abusers, drug abusers and alcoholics;
6. Allergic to lenvatinib or other treatments.
7. Severe mental or nervous system disorders affecting informed consent and / or expression or observation of adverse reaction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
MST | 24 months
  Median Survival Time (MST) was defined as the duration from the date of patient recruited to the date of death from any cause

SECONDARY OUTCOMES:
ORR | Assessment in 1 to 3 months after radiotherapy
  Overall Response Rate (ORR) was defined as the total of CR (Complete Response) and PR (Partial Response). CR and PR were assessed by independent reviewers according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. ORR evaluated in 1 to 3 months after the completion of radiotherapy.
TTP | 24 months
  Time to Progression (TTP) was defined as the duration from the date of patient recruited to the first progress at any site or the date of death
Rate of III-IV grade adverse events | up to 24 months
  Adverse events was evaluated during received protocol therapy according to CTCAE 4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Bo Chen, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No